CLINICAL TRIAL: NCT00687323
Title: Phase II Study of Temozolomide in Previously Untreated Acute Myeloid Leukemia (AML)/Myelodysplastic Syndrome (MDS) Subjects Unsuitable for Standard Induction Therapy Exhibiting Low MGMT Expression
Brief Title: Study of Temozolomide in Previously Untreated Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS) Participants With Low O6-Methylguanine Methyltransferase (MGMT) Expression (P05052)
Acronym: TALL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05052; MK-7365-240
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Results first posted 2012-07-18 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-05

CONDITIONS: Leukemia, Acute Myeloid; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Temozolomide (Experimental): Temozolomide capsules orally, once daily: 1 induction cycle (200 mg/m^2/day for 7 days in 1 28 day cycle), 1 consolidation cycle (200 mg/m^2/day for 7 days in 1 28 day cycle), then 200 mg/m^2/day for 7 days each 28-day cycle or for 5 days each 28-day cycle (12 cycle maximum). Alternatively participants could have received 100 mg/m^2/day for 21 days of each 28-day cycle (12 cycle maximum).
  Interventions: Drug: temozolomide

INTERVENTIONS:
Drug: temozolomide
  Other Names: Temodol; SCH 052365; MK-7365

SUMMARY:
The primary objective of this study is to evaluate the safety, tolerability, and efficacy of temozolomide in acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS) participants who are not candidates for standard induction therapy and exhibit low MGMT expression.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of acute myeloid leukemia (AML), any subtype except acute promyelocytic leukemia (APL), by the World Health Organization (WHO) criteria, or high risk MDS with blasts between 10 and 20% in the bone marrow.
* No prior AML chemotherapy except hydroxyurea.
* Leukemic blast count <30x10^9/L at the start of therapy. Prior cytoreduction with hydroxyurea (maximum 14 days) is permitted.
* Participant is not a candidate for aggressive induction based on at least one of the following: adverse-risk cytogenetics (complete or partial deletion of 5 or 7, complex [>3] cytogenetic abnormalities, inv3, 11q23 abnormalities); secondary AML (antecedent hematologic disorder or therapy-related AML); comorbid medical illnesses precluding standard induction therapy; participant's refusal of standard induction therapy.
* Confirmed low MGMT expression (MGMT: beta-actin ≤0.2), as evaluated by Western blot, or weak MGMT expression defined as > 0.2 and ≤2.5 if promoter is methylated, upon Sponsor approval.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Use of medically approved contraception in fertile males and females.
* Negative urine or serum pregnancy test for women of childbearing potential (72 hours prior to Baseline).

Exclusion Criteria:

* Serum bilirubin >2 times the upper limit of normal (ULN), or serum aspartate aminotransferase/ alanine aminotransferase >5 times ULN.
* Serum creatinine >200 umol/L.
* History of other malignancies within 1 year prior to study entry, with the exception of localized nonmelanomatous skin cancer or cervical cancer in situ.
* Presence of active uncontrolled infection.
* Known human immunodeficiency virus (HIV) infection.
* Any medical condition that may interfere with protocol evaluation or oral medication intake.
* Prior chemotherapy other than hydroxyurea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2007-07-30 (Actual); Primary Completion 2011-05-09 (Actual); Study Completion 2012-12-23 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Brandwein JM, Yang L, Schimmer AD, Schuh AC, Gupta V, Wells RA, Alibhai SM, Xu W, Minden MD. A phase II study of temozolomide therapy for poor-risk patients aged >or=60 years with acute myeloid leukemia: low levels of MGMT predict for response. Leukemia. 2007 Apr;21(4):821-4. doi: 10.1038/sj.leu.2404545. Epub 2007 Jan 25. No abstract available. PMID 17252015

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Temozolomide
Started | 195 (Number of screened participants)
Received Treatment | 47
Completed | 15 (Number of participants alive at one year)
Not Completed | 180
Not completed — Death | 25
Not completed — Withdrawal by Subject | 1
Not completed — Excluded from efficacy evaluations | 6
Not completed — Screen failure | 148

BASELINE CHARACTERISTICS:
Arm/Group | Temozolomide
Number analyzed (Participants) | 47
Age, Continuous [Mean (Full Range); unit: years] — Number of participants who received treatment
  years | 75 [52 to 89]
Sex: Female, Male [Count of Participants; unit: Participants] — Number of participants who received treatment
  Participants
    Female | 18
    Male | 29
Region of Enrollment [Number; unit: participants] — Number of participants who received treatment
  participants
    Canada | 47

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response at the End of Temozolomide Induction
Description: Complete Response (CR): < 5% blasts in normocellular bone marrow (BM); Absolute Neutrophil Count (ANC) > 1.0 x 10^9/L, platelets > 100 x 10^9/L, and no extramedullary disease.
  CR with incomplete platelet recovery (CRp): All the criteria of CR but with platelets < 100 x 10^9/L but ≥ 50 x 10^9/L and platelet transfusion independent.
  Morphologic leukemia-free state (MLFS): complete clearance of blasts from marrow and blood, but criteria for CR or CRp not met.
  Partial response (PR): decrease ≥ 50% BM blasts. Minimal Response (MR): decrease ≥ 25% but <50% BM blasts.
Time Frame: at the end of each cycle (approximately 4 weeks post start of cycle), up to a maximum 63 weeks
Population: Efficacy evaluable population (all eligible participants who completed at least one additional disease evaluation after baseline)
Measure: Number; unit: participants
Arm/Group | Temozolomide
Number analyzed (Participants) | 41
participants
  CR | 10
  CRp | 2
  MLFS | 4
  PR | 8
  MR | 7

2. Secondary Outcome: Duration of Response in Participants Achieving Complete Response (CR) and Proceeding to Reduced Dose-intensity Maintenance Therapy With Temozolomide
Description: Complete Response (CR): < 5% blasts in normocellular bone marrow (BM); Absolute Neutrophil Count (ANC) > 1.0 x 10^9/L, platelets > 100 x 10^9/L, and no extramedullary disease.
Time Frame: Up to 1 year after treatment ends (up to 115 weeks)
Population: as for outcome 1
Measure: Median (Full Range); unit: Days
Arm/Group | Temozolomide
Number analyzed (Participants) | 41
Days | 408 [101 to 946]

3. Secondary Outcome: Relapse-free Survival in Participants Achieving CR or CRp and Proceeding to Reduced Dose-intensity Maintenance Therapy With Temozolomide
Description: Relapse-free survival was defined as time to disease progression. Complete Response (CR): < 5% blasts in normocellular bone marrow (BM); Absolute Neutrophil Count (ANC) > 1.0 x 10^9/L, platelets > 100 x 10^9/L, and no extramedullary disease. CR with incomplete platelet recovery (CRp): All the criteria of CR but with platelets < 100 x 10^9/L but ≥ 50 x 10^9/L and platelet transfusion independent.
Time Frame: Start of treatment until disease progression [up to 1 year after treatment ends (up to 115 weeks)]
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temozolomide
Number analyzed (Participants) | 41
months | 10.5 [4.2 to 19.5]

4. Secondary Outcome: Overall Survival (OS) in Participants Achieving CR or CRp and Proceeding to Reduced Dose-intensity Maintenance Therapy With Temozolomide
Description: OS was defined as the time from start of treatment until death or end of study.
  Complete Response (CR): < 5% blasts in normocellular bone marrow (BM); Absolute Neutrophil Count (ANC) > 1.0 x 10^9/L, platelets > 100 x 10^9/L, and no extramedullary disease. CR with incomplete platelet recovery (CRp): All the criteria of CR but with platelets < 100 x 10^9/L but ≥ 50 x 10^9/L and platelet transfusion independent.
Time Frame: Start of treatment until death or end of study [up to 1 year after treatment ends (up to 115 weeks)]
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temozolomide
Number analyzed (Participants) | 41
months | 21.4 [9.7 to NA] — not achieved

5. Secondary Outcome: Number of Previously Untreated Participants With Low O6-Methylguanine Methyltransferase (MGMT) Expression
Description: Low MGMT expression was defined as MGMT/β-actin ratio < 0.2. MGMT & β-actin are cancer biomarkers.
Time Frame: Baseline
Population: All screened participants
Measure: Number; unit: participants
Arm/Group | Temozolomide
Number analyzed (Participants) | 195
participants | 81

6. Secondary Outcome: MGMT Expression in Leukemic Blasts at the Time of Relapse
Description: Low MGMT expression was defined as MGMT/β-actin ratio of <0.2.
  MGMT & β-actin are cancer biomarkers.
Time Frame: Up to 1 year after treatment ends (up to 115 weeks)
Population: Analysis could not be performed due to lack of specimens.
Arm/Group | Temozolomide
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants With CR, PR, or MLFS Who Received Modified Low Dose Maintenance Therapy (100 mg/m^2/Day x21 Days of Each 28 Day Cycle) and Experienced Toxicity
Description: Toxicity was defined as any adverse event experienced by a participant regardless of causal relationship with study treatment. An adverse event (AE) was defined as any untoward medical occurrence in a participant administered a pharmaceutical product, biologic (at any dose), or medical device, which did not necessarily have a causal relationship with the treatment. Adverse events may have included the onset of new illness and/or the exacerbation of preexisting conditions.
Time Frame: From first dose to 30 days after last dose of study drug (up to 67 weeks)
Population: Number of participants who achieved CR, PR, or MLFS and received modified low dose maintenance therapy
Measure: Number; unit: participants
Arm/Group | Temozolomide
Number analyzed (Participants) | 1
participants | 1

8. Secondary Outcome: Progression-free Survival for Participants Achieving PR, MLSF, or MR
Description: Progression-free survival was defined as time to disease progression. Morphologic leukemia-free state (MLFS): complete clearance of blasts from marrow and blood, but criteria for CR or CRp not met. Partial response (PR): decrease ≥ 50% BM blasts. Minimal Response (MR): decrease ≥ 25% but <50% BM blasts.
Time Frame: Start of treatment until disease progression [up to 1 year after treatment ends (up to 115 weeks)]
Population: Efficacy evaluable population (all eligible participants who completed at least one additional disease evaluation after baseline) who achieved PR, MLSF, or MR
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temozolomide
Number analyzed (Participants) | 19
months | 1.6 [0.3 to 5.8]

9. Secondary Outcome: Quality of Life (QoL) in Participants Receiving Long Term Temozolomide Therapy Assessed by European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-30
Description: The EORTC QLQ-C30 was a 30-item questionnaire developed to assess the QoL of cancer patients. Scores ranged from 0 -100. For functional and global QoL scales, higher scores meant a better level of function. For symptom-oriented scales, a higher score meant more severe symptoms and a decrease in QoL.
Time Frame: Baseline and post-study visit (63 weeks)
Population: Analysis could not be performed due to incomplete data.
Arm/Group | Temozolomide
Number analyzed (Participants) | 0

10. Secondary Outcome: Quality of Life (QoL) in Participants Receiving Long Term Temozolomide Therapy Assessed by EORTC QLQ-LC13
Description: The EORTC QLQ-LC13 was a 13-item questionnaire developed to supplement the EORTC QLQ-C30 in lung cancer patients. It had a score range 0-100 with higher scores representing an increase in symptoms.
Time Frame: Baseline and post-study visit (63 weeks)
Population: Analysis could not be performed due to incomplete data.
Arm/Group | Temozolomide
Number analyzed (Participants) | 0

11. Secondary Outcome: Quality of Life (QoL) in Participants Receiving Long Term Temozolomide Therapy Assessed by Functional Assessment of Cancer Therapy (FACT)-G
Description: The FACT-G was a 27-item questionnaire developed to assess the QoL in patients with chronic illnesses. Scores ranged from 0 to 28. For physical well being, lower scores indicated a better outcome. For functional well being, higher scores indicated a better outcome. For social & emotional well being, whether a high score or a lower one indicated a better outcome depended on the question.
Time Frame: Baseline and post-study visit (63 weeks)
Population: Analysis could not be performed due to incomplete data.
Arm/Group | Temozolomide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Population was all treated participants.
Arm/Group | TEMOZOLOMIDE
Serious Adverse Events (participants affected / at risk) | 25/47
Other Adverse Events (participants affected / at risk) | 45/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TEMOZOLOMIDE (N=47)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 5 (6)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
NEUTROPHILIA (Blood and lymphatic system disorders) | 1 (1)
COLONIC STENOSIS (Gastrointestinal disorders) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 3 (3)
MELAENA (Gastrointestinal disorders) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 2 (2)
VOMITING (Gastrointestinal disorders) | 1 (1)
ASTHENIA (General disorders) | 2 (2)
FATIGUE (General disorders) | 2 (2)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 2 (2)
HYPERTHERMIA (General disorders) | 1 (1)
MUCOSAL INFLAMMATION (General disorders) | 1 (1)
PYREXIA (General disorders) | 2 (2)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1)
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 1 (1)
CYSTITIS (Infections and infestations) | 1 (1)
DIVERTICULITIS (Infections and infestations) | 1 (1)
FUNGAL INFECTION (Infections and infestations) | 1 (1)
GASTROINTESTINAL FUNGAL INFECTION (Infections and infestations) | 1 (1)
HERPES SIMPLEX (Infections and infestations) | 1 (1)
INFECTION (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 7 (7)
PNEUMONIA RESPIRATORY SYNCYTIAL VIRAL (Infections and infestations) | 1 (1)
PSEUDOMONAL SEPSIS (Infections and infestations) | 1 (1)
PYOMYOSITIS (Infections and infestations) | 1 (1)
SEPSIS (Infections and infestations) | 3 (3)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 2 (2)
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 (2)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 1 (1)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 (1)
SYNCOPE (Nervous system disorders) | 2 (2)
RENAL FAILURE (Renal and urinary disorders) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4 (4)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
HYPOTENSION (Vascular disorders) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1)
NEUTROPENIC INFECTION (Infections and infestations) | 1 (1)
PNEUMONIA FUNGAL (Infections and infestations) | 1 (1)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TEMOZOLOMIDE (N=47)
ANAEMIA (Blood and lymphatic system disorders) | 6 (6)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 8 (9)
NEUTROPENIA (Blood and lymphatic system disorders) | 4 (4)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 7 (8)
CONSTIPATION (Gastrointestinal disorders) | 16 (34)
DIARRHOEA (Gastrointestinal disorders) | 6 (7)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 3 (3)
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 5 (5)
NAUSEA (Gastrointestinal disorders) | 14 (25)
STOMATITIS (Gastrointestinal disorders) | 3 (3)
VOMITING (Gastrointestinal disorders) | 9 (12)
ASTHENIA (General disorders) | 6 (6)
CHILLS (General disorders) | 5 (5)
FATIGUE (General disorders) | 26 (34)
HYPERTHERMIA (General disorders) | 4 (4)
MUCOSAL INFLAMMATION (General disorders) | 3 (3)
OEDEMA (General disorders) | 4 (5)
OEDEMA PERIPHERAL (General disorders) | 5 (5)
PYREXIA (General disorders) | 10 (13)
NASOPHARYNGITIS (Infections and infestations) | 3 (3)
ORAL HERPES (Infections and infestations) | 3 (3)
URINARY TRACT INFECTION (Infections and infestations) | 5 (5)
CONTUSION (Injury, poisoning and procedural complications) | 6 (8)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 (4)
BLOOD CREATININE INCREASED (Investigations) | 3 (3)
HAEMOGLOBIN DECREASED (Investigations) | 4 (4)
PLATELET COUNT DECREASED (Investigations) | 3 (5)
WEIGHT DECREASED (Investigations) | 3 (3)
DECREASED APPETITE (Metabolism and nutrition disorders) | 19 (22)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 8 (8)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 5 (7)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 (6)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 (5)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 3 (3)
DIZZINESS (Nervous system disorders) | 5 (5)
DYSGEUSIA (Nervous system disorders) | 4 (5)
HEADACHE (Nervous system disorders) | 6 (8)
CONFUSIONAL STATE (Psychiatric disorders) | 5 (5)
INSOMNIA (Psychiatric disorders) | 4 (4)
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 (5)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 10 (12)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3 (3)
DRY SKIN (Skin and subcutaneous tissue disorders) | 4 (4)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 4 (6)
PETECHIAE (Skin and subcutaneous tissue disorders) | 10 (10)
RASH (Skin and subcutaneous tissue disorders) | 7 (9)
HYPOTENSION (Vascular disorders) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study Chair agrees not to publish/present any interim results without the Sponsor's prior written consent. The Principal Investigators (PIs) agree to provide 30 days prior to submission to the Sponsor to review copies of abstracts/manuscripts. The Sponsor shall have proper representation on publications and editorial rights with regard to data analysis, presentation, proprietary information, and accuracy. If the parties disagree, the PIs agree to meet with the Sponsor to discuss/resolve.